CLINICAL TRIAL: NCT03579693
Title: Cross-over Randomized Controlled Trial of Coenzyme Q10 or Nicotinamide Riboside in Chronic Kidney Disease
Brief Title: Trial of Nicotinamide Riboside and Co-enzyme Q10 in Chronic Kidney Disease
Acronym: CoNR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Bryan Kestenbaum, Professor, School of Medicine: Department of Medicine: Nephrology, University of Washington
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00004998; R01DK101509 (NIH)
Record Dates: First submitted 2018-06-25; First posted 2018-07-06 (Actual); Results first posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-12

CONDITIONS: Chronic Kidney Disease; Sarcopenia; Frailty
Keywords: Mitochondria; Antioxidants; CoQ10; Nicotinamide riboside; Ergometry; Fatigue; Aerobic capacity
MeSH Terms: conditions — Renal Insufficiency, Chronic; Sarcopenia; Frailty; Fatigue | interventions — coenzyme Q10; nicotinamide-beta-riboside

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, cross-over trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- CoQ10 (Active Comparator): Coenzyme Q10, 2 - 250 mg tablets twice a day (1000 mg total daily dose) for 6 weeks
  Interventions: Dietary Supplement: CoQ10
- Nicotinamide riboside (Active Comparator): Nicotinamide riboside, 1 - 600 mg tablet twice a day (1200 mg total daily dose) for 6 weeks
  Interventions: Dietary Supplement: Nicotinamide riboside
- Placebo (Placebo Comparator): Placebo, inactive sugar pill for 6 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: CoQ10 — CoQ10 tablet
  Other Names: coenzyme Q10
  Arms: CoQ10
Dietary Supplement: Nicotinamide riboside — NR tablet
  Other Names: NR
  Arms: Nicotinamide riboside
Dietary Supplement: Placebo — Sugar pill designed to mimic coQ10 and NR
  Arms: Placebo

SUMMARY:
Chronic kidney disease is associated with the loss of skeletal muscle mass and function. This process detrimentally impacts mobility, functional independence, and quality of life. Mounting evidence suggests that chronic kidney disease impairs skeletal muscle functioning by injuring mitochondria, the central energy producing units of cells.

Potential treatment options to restore mitochondrial function include aerobic and weight bearing exercise and medications that directly improve mitochondrial energetics. Unfortunately, exercise programs may be difficult to implement in people who have chronic diseases, such as kidney disease.. Coenzyme Q10 (coQ10) and nicotinamide riboside (NR) are naturally occurring supplements that can directly improve mitochondrial efficiency. Both compounds help mitochondria produce more energy while generating less waste.

The primary purpose of this study is to test whether coQ10 and NR can improve muscle function among people with chronic kidney disease. What we learn in this study may help us better understand the mechanisms of skeletal muscle impairment among people with kidney disease and ultimately improve their ability to be active and independent.

DETAILED DESCRIPTION:
Sarcopenia (decreased muscle mass or function) is common in patients with chronic kidney disease (CKD) patients with direct impacts on their metabolic and clinical outcomes. Existing evidence and the investigator's preliminary data suggest that mitochondrial dysfunction is a key underlying mechanism of sarcopenia in CKD. However, the ability of treatments to modify mitochondrial functioning in CKD patients is unknown. Coenzyme Q10 (coQ10) and nicotinamide riboside (NR) are naturally occurring supplements that reduce oxidative stress and restore substrate delivery to mitochondria, respectively.

Both processes have the potential to increase mitochondrial energy production with direct consequences for many metabolic and physical processes, including:

* aerobic capacity
* work efficiency
* mitochondrial energetics
* fatigue
* physical function
* inflammation
* oxidative stress
* heart failure symptoms
* metabolomics

These outcomes will assessed in all study participants who enroll in the trial. Addressing these knowledge gaps is necessary to shed new light on the pathophysiology of sarcopenia in CKD and suggest future interventions that reduce morbidity and mortality.

This is a randomized, placebo-controlled, double-blind crossover trial of coQ10 and NR treatments. Participants will receive coQ10 (1000 mg daily), NR (1200 mg daily), or placebo each for six-weeks in random order with a 7-day washout between treatment periods. The primary outcomes are aerobic capacity and muscle work efficiency, measured during cycle ergometry.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease, defined in this study as an estimated glomerular filtration rate (eGFR) of <50ml/min/1.73m2 using the Chronic Kidney Disease Epidemiology Collaboration equation

Exclusion Criteria:

* 6-minute walking distance >500meters
* Pregnancy
* Receiving renal replacement therapy (dialysis or kidney transplantation)
* Expectation to start dialysis within 6 months
* Insulin dependent diabetes mellitus
* Severe anemia: hemoglobin <8 g/dL
* Hyperkalemia: K >5.7 mEq/L
* Weight >300 lbs
* HIV
* End stage liver disease with cirrhosis
* Oxygen-dependent Chronic Obstructive Pulmonary Disease (COPD)
* Unable to walk unassisted from room to room in own house
* Institutionalization, or inability to consent
* Use of immunosuppressive medications (i.e. steroids, calcineurin inhibitors)
* Malignancy requiring active treatment or currently under surveillance (at the discretion of the investigator)
* Cardiac pacemaker
* Current participation in another interventional trial
* Non-English speaking
* Hospitalization for heart attack, stroke, or unstable cardiac chest pain within the previous 3 months (e.g. myocardial infarction, unstable angina, cerebrovascular accident)
* Any medical condition that the investigator feels would prevent the participant from safely completing the exercise-based outcome measurements.
* Baseline systolic blood pressure >170 or diastolic blood pressure >100
* Persistent or permanent uncontrolled arrhythmia (at the discretion of the investigator)

Ages: 30 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Kestenbaum, MD, Principal Investigator — University of Washington; Baback Roshanravan, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ahmadi A, Valencia AP, Begue G, Norman JE, Fan S, Durbin-Johnson BP, Jenner BN, Campbell MD, Reyes G, Kapahi P, Himmelfarb J, de Boer IH, Marcinek DJ, Kestenbaum BR, Gamboa JL, Roshanravan B. A Pilot Trial of Nicotinamide Riboside and Coenzyme Q10 on Inflammation and Oxidative Stress in CKD. Clin J Am Soc Nephrol. 2025 Mar 1;20(3):346-357. doi: 10.2215/CJN.0000000624. Epub 2025 Jan 23. PMID 39847432
- [Derived] Ahmadi A, Begue G, Valencia AP, Norman JE, Lidgard B, Bennett BJ, Van Doren MP, Marcinek DJ, Fan S, Prince DK, Gamboa J, Himmelfarb J, de Boer IH, Kestenbaum BR, Roshanravan B. Randomized crossover clinical trial of coenzyme Q10 and nicotinamide riboside in chronic kidney disease. JCI Insight. 2023 Jun 8;8(11):e167274. doi: 10.1172/jci.insight.167274. PMID 37159264
- See also: Website for the Kidney Research Institute at the University of Washington — https://kri.washington.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo, Then Nicotinamide Riboside, Then CoQ10: Placebo, inactive sugar pill for 6 weeks; then washout for 1 week; then nicotinamide riboside, 1 - 600 mg tablet twice a day (1200 mg total daily dose) for 6 weeks; then washout for 1 week; then coenzyme Q10, 2 - 250 mg tablets twice a day (1000 mg total daily dose) for 6 weeks.
- Placebo, Then CoQ10, Then Nicotinamide Riboside: Placebo, inactive sugar pill for 6 weeks; then washout for 1 week; then coenzyme Q10, 2 - 250 mg tablets twice a day (1000 mg total daily dose) for 6 weeks; then washout for 1 week; then nicotinamide riboside, 1 - 600 mg tablet twice a day (1200 mg total daily dose) for 6 weeks.
- Nicotinamide Riboside, Then Placebo, Then CoQ10: Nicotinamide riboside, 1 - 600 mg tablet twice a day (1200 mg total daily dose) for 6 weeks; then washout for 1 week; placebo, inactive sugar pill for 6 weeks; then washout for 1 week; then coenzyme Q10, 2 - 250 mg tablets twice a day (1000 mg total daily dose) for 6 weeks.
- Nicotinamide Riboside, Then CoQ10, Then Placebo: Nicotinamide riboside, 1 - 600 mg tablet twice a day (1200 mg total daily dose) for 6 weeks; then washout for 1 week; then coenzyme Q10, 2 - 250 mg tablets twice a day (1000 mg total daily dose) for 6 weeks; then washout for 1 week; placebo, inactive sugar pill for 6 weeks.
- CoQ10, Then Placebo, Then Nicotinamide Riboside: Coenzyme Q10, 2 - 250 mg tablets twice a day (1000 mg total daily dose) for 6 weeks; then washout for 1 week; then placebo, inactive sugar pill for 6 weeks; then washout for 1 week; then nicotinamide riboside, 1 - 600 mg tablet twice a day (1200 mg total daily dose) for 6 weeks.
- CoQ10, Then Nicotinamide Riboside, Then Placebo: Coenzyme Q10, 2 - 250 mg tablets twice a day (1000 mg total daily dose) for 6 weeks; then washout for 1 week; then nicotinamide riboside, 1 - 600 mg tablet twice a day (1200 mg total daily dose) for 6 weeks; then washout for 1 week; then placebo, inactive sugar pill for 6 weeks.
Period: First Intervention (6 Weeks)
Arm/Group | Placebo, Then Nicotinamide Riboside, Then CoQ10 | Placebo, Then CoQ10, Then Nicotinamide Riboside | Nicotinamide Riboside, Then Placebo, Then CoQ10 | Nicotinamide Riboside, Then CoQ10, Then Placebo | CoQ10, Then Placebo, Then Nicotinamide Riboside | CoQ10, Then Nicotinamide Riboside, Then Placebo
Started | 4 | 5 | 5 | 4 | 4 | 4
Completed | 4 | 5 | 5 | 4 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Period: Washout (1 Week)
Arm/Group | Placebo, Then Nicotinamide Riboside, Then CoQ10 | Placebo, Then CoQ10, Then Nicotinamide Riboside | Nicotinamide Riboside, Then Placebo, Then CoQ10 | Nicotinamide Riboside, Then CoQ10, Then Placebo | CoQ10, Then Placebo, Then Nicotinamide Riboside | CoQ10, Then Nicotinamide Riboside, Then Placebo
Started | 4 | 5 | 5 | 4 | 4 | 3
Completed | 4 | 5 | 5 | 4 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention (6 Weeks)
Arm/Group | Placebo, Then Nicotinamide Riboside, Then CoQ10 | Placebo, Then CoQ10, Then Nicotinamide Riboside | Nicotinamide Riboside, Then Placebo, Then CoQ10 | Nicotinamide Riboside, Then CoQ10, Then Placebo | CoQ10, Then Placebo, Then Nicotinamide Riboside | CoQ10, Then Nicotinamide Riboside, Then Placebo
Started | 4 | 5 | 5 | 4 | 4 | 3
Completed | 4 | 4 | 5 | 4 | 4 | 3
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Period: Second Washout (1 Week)
Arm/Group | Placebo, Then Nicotinamide Riboside, Then CoQ10 | Placebo, Then CoQ10, Then Nicotinamide Riboside | Nicotinamide Riboside, Then Placebo, Then CoQ10 | Nicotinamide Riboside, Then CoQ10, Then Placebo | CoQ10, Then Placebo, Then Nicotinamide Riboside | CoQ10, Then Nicotinamide Riboside, Then Placebo
Started | 4 | 5 | 5 | 4 | 4 | 3
Completed | 4 | 5 | 5 | 4 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention (6 Weeks)
Arm/Group | Placebo, Then Nicotinamide Riboside, Then CoQ10 | Placebo, Then CoQ10, Then Nicotinamide Riboside | Nicotinamide Riboside, Then Placebo, Then CoQ10 | Nicotinamide Riboside, Then CoQ10, Then Placebo | CoQ10, Then Placebo, Then Nicotinamide Riboside | CoQ10, Then Nicotinamide Riboside, Then Placebo
Started | 4 | 5 | 5 | 4 | 4 | 3
Completed | 4 | 5 | 5 | 4 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo, Then Nicotinamide Riboside, Then CoQ10 | Placebo, Then CoQ10, Then Nicotinamide Riboside | Nicotinamide Riboside, Then Placebo, Then CoQ10 | Nicotinamide Riboside, Then CoQ10, Then Placebo | CoQ10, Then Placebo, Then Nicotinamide Riboside | CoQ10, Then Nicotinamide Riboside, Then Placebo | Total
Number analyzed (Participants) | 4 | 5 | 5 | 4 | 4 | 4 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (3.0) | 63.4 (11.8) | 63.6 (4.8) | 56.2 (16.3) | 64.0 (7.5) | 58.2 (22.6) | 61.5 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 2 | 0 | 3 | 4 | 16
  Male | 0 | 2 | 3 | 4 | 1 | 0 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 4 | 5 | 5 | 4 | 4 | 3 | 25
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 0 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 1
  White | 4 | 5 | 3 | 4 | 1 | 4 | 21
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 5 | 5 | 4 | 4 | 4 | 26
eGFR per 2021 CKD-EPI [Mean (Standard Deviation); unit: mL/min/1.73m^2] | 33.6 (10.5) | 39.3 (10.1) | 32.6 (7.8) | 34.6 (10.5) | 45.2 (8.0) | 36.0 (4.5) | 37.0 (9.0)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 27.9 (7.9) | 27.9 (4.8) | 29.6 (4.0) | 25.3 (4.6) | 25.8 (2.7) | 29.9 (8.4) | 27.7 (5.2)

OUTCOME MEASURES:

1. Primary Outcome: Maximal Aerobic Capacity- CoQ10
Description: The maximal aerobic capacity (oxygen uptake mL/min/kg body weight) during cycle ergometry at the end of each treatment period.
Time Frame: 6 weeks
Population: Randomized participants that completed cycle ergometry following each treatment period.
Measure: Mean (Standard Deviation); unit: mL/min/kg
Arm/Group | CoQ10 | Nicotinamide Riboside | Placebo
Number analyzed (Participants) | 24 | 25 | 25
mL/min/kg | 21.4 (4.7) | 20.7 (4.7) | 20.7 (4.8)
Statistical Analysis 1: Comparison: CoQ10 vs Placebo; Test type: Superiority; p = 0.33, Mixed Models Analysis; Mean Difference (Final Values) = 0.44, 95% CI 2-sided [-0.43 to 1.31] — Interpretation of mean difference is for a typical participant, i.e. random effect of 0
Statistical Analysis 2: Comparison: Nicotinamide Riboside vs Placebo; Test type: Superiority; p = 0.93, Mixed Models Analysis; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.90 to 0.82] — Interpretation of mean difference is for a typical participant, i.e. random effect of 0

2. Primary Outcome: Work Efficiency
Description: The work efficiency (oxygen uptake mL/min/kg body weight at a specified constant of 60 watts work rate for 3 minutes) during cycle ergometry at the end of each treatment period. This is reported as the work performed at 60 watts divided by the energy expended at 0 watts times 100, and reported on the percent scale..
Time Frame: 6 weeks
Population: Includes participants randomized and treated who complete cycle ergometry at the end of the corresponding treatment period.
Measure: Mean (Standard Deviation); unit: Percent difference
Arm/Group | CoQ10 | Nicotinamide Riboside | Placebo
Number analyzed (Participants) | 24 | 25 | 25
Percent difference | 33.3 (4.2) | 32.5 (5.1) | 33.1 (5.2)
Statistical Analysis 1: Comparison: CoQ10 vs Placebo; Test type: Superiority; p = 0.050, Mixed Models Analysis; Mean Difference (Final Values) = -1.76, 95% CI 2-sided [-3.47 to 0.00] — Interpretation of mean difference is for a typical participant, i.e. random effect of 0
Statistical Analysis 2: Comparison: Nicotinamide Riboside vs Placebo; Test type: Superiority; p = 0.47, Mixed Models Analysis; Mean Difference (Final Values) = -0.62, 95% CI 2-sided [-2.28 to 1.05] — Interpretation of mean difference is for a typical participant, i.e. random effect of 0

ADVERSE EVENTS:
Time Frame: For each treatment arm, adverse events are reported from the start of the treatment until the next visit (approximately 6 weeks total for each treatment).
Description: Definitions used were consistent with clinicaltrials.gov. At each visit potential adverse events were assessed by participant interview.
Arm/Group | CoQ10 | Nicotinamide Riboside | Placebo
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 1/25 | 2/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CoQ10 (N=25) | Nicotinamide Riboside (N=25) | Placebo (N=25)
Upper respiratory illness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-08): https://cdn.clinicaltrials.gov/large-docs/93/NCT03579693/Prot_SAP_001.pdf